CLINICAL TRIAL: NCT07130266
Title: Evaluation of the Clinical and Volumetric Effectiveness of 0.8% Hyaluronic Acid Gel Adjunct to Open-Flap Surgery in Periodontitis Patients With Thin Gingival Phenotype
Brief Title: Adjunctive 0.8% Hyaluronic Acid Gel in Open-Flap Surgery for Thin Gingival Phenotype in Patients With Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E.69156; 20220801 (Other Grant/Funding Number: Bezmialem Vakif University)
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Hyaluronic Acid; Open Flap Debridement; Periodontitis; Gingival Phenotype; Gingival Recession
Keywords: Hyaluronic acid; Periodontitis; Open Flap Debridement; Gingival recession
MeSH Terms: conditions — Periodontitis; Gingival Recession

STUDY DESIGN:
Intervention Model Description: During the surgery session, patients were block randomized, with the allocation order using a computer program (www.randomizer.org.). Group assignment was carried out by another investigator who was not involved in the treatment procedure or clinical measurements (UGE). Study groups were as follows:
  1. OFD + 0.8% HA gel (n = 20, test group)
  2. OFD alone (n = 20, control group).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open Flap Debridement (OFD) (Placebo Comparator): Open flap debridement was carried out, and the surgical site was irrigated with physiological saline in a manner consistent with the HA gel application protocol in the test group. A second application of physiological saline to the sulcus area was performed four weeks postoperatively
  Interventions: Procedure: giving an impression of the application
- Open Flap Debridement (OFD)+HA (Active Comparator): Open flap debridement was carried out, and 1 ml of 0.8% HA gel was applied to the root surfaces of the affected teeth, bone, and the inner surface of the flap in the surgical area for 2 minutes. HA gel application was repeated at four weeks postoperatively.
  Interventions: Procedure: Procedure/Surgery: Hyaluronic acid gel application

INTERVENTIONS:
Procedure: Procedure/Surgery: Hyaluronic acid gel application — After root surface cleaning and infected cement removal, 0.8% HA gel was applied to the root surface, bone, and inner surface of the flap and left for 2 minutes.
  Arms: Open Flap Debridement (OFD)+HA
Procedure: giving an impression of the application — In the control group, instead of HA gel, the area was irrigated with physiological saline solution.
  Arms: Open Flap Debridement (OFD)

SUMMARY:
The aim of this study is to evaluate the clinical effectiveness of 0.8% hyaluronic acid (HA) gel as an adjunct to open flap debridement (OFD) in periodontitis patients with a thin gingival phenotype.

The primary research question is:

Does the adjunctive use of 0.8% HA gel reduce gingival recession and improve clinical parameters? To answer this, researchers will compare the adjunctive use of 0.8% HA gel to physiological saline in combination with OFD, assessing their effects on clinical outcomes and gingival recession in patients with a thin gingival phenotype.

Participants will:

* Receive 0.8% HA gel application during OFD surgery and a second application at 4 weeks postoperatively.
* Attend follow-up visits at 1, 3, and 6 months after surgery for clinical assessments and measurements.

DETAILED DESCRIPTION:
A total of 40 patients were enrolled in the study and randomly assigned to two groups: (a) OFD + 0.8% HA gel (n = 20, test group) and (b) OFD alone (n = 20, control group). Clinical parameters including plaque (P), bleeding on probing (BoP), probing pocket depth (PPD), and clinical attachment level (CAL) were recorded at baseline. Following initial periodontal therapy, sites with PPD ≥ 5 mm and horizontal bone loss, were identified in patients with a thin gingival phenotype, determined using color-coded gingival probes. Intraoral digital scans were taken, and relative gingival recession (rGR) was recorded immediately before surgery.

During OFD, the test group received adjunctive 0.8% HA gel, while the control group received physiological saline. In the test group, HA gel application was repeated at 4 weeks postoperatively. Changes in soft tissue volume (mm³) and thickness (mm) were measured using specialized computer software. Follow-up evaluations were performed at 3 and 6 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of periodontitis (Stage II/III);
2. Presence of horizontal bone loss with at least three adjacent teeth, each exhibiting a probing depth ≥ 5mm and a keratinized tissue width ≥ 2mm on single-rooted teeth;
3. a thin gingival phenotype;
4. Areas with horizontal bone loss without intra-bony defects, where no additional hard and soft tissue augmentation was required
5. a full-mouth plaque score (FMPS) and full-mouth bleeding score (FMBS <20%.

Exclusion Criteria:

* Systemic diseases
* Smokers
* Pregnant or lactating women
* Those who received periodontal treatment within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level (CAL) | Baseline - 3months - 6 months
  CAL were measured from both the buccal and palatal/lingual aspects of each tooth at six points including mesial, distal, and midpoint, and recorded in mm. CAL was measured as the distance between the base of the pocket and the enamel cement junction.

SECONDARY OUTCOMES:
3D Measurements | Baseline - 3months - 6 months
  The median tooth in the area of three adjacent teeth undergoing surgery was chosen for analysis, as it included the interproximal papilla regions of the adjacent teeth treated with periodontal surgery. Data from the 3rd and 6th months intraoral digital scans were extracted separately from the baseline, and the region for volumetric analysis was divided into three equal parts: mesial, distal, and middle. The interproximal and middle regions were evaluated separately, and the volumetric changes over time were calculated in mm³ using the program.
Analysis of 2D Gingival Thickness Changes | Baseline - 3months - 6 months
  The change in gingival thickness at all time points was calculated using standard reference points on the previously superimposed models. Gingival thickness change was measured in 2D at these points, and repeated for both buccal and palatal/lingual regions.
Relative gingival recession (rGR) | Baseline - 3months - 6 months
  The distance between the horizontal reference point on the acrylic stent and the marginal gingiva at the surgical site was measured and recorded as relative gingival recession (rGR).
Probing depth (PD) | Baseline - 3months - 6 months
  Defined as the distance from the base of the periodontal pocket to the marginal gingiva
Plaque (P) | Baseline - 3months - 6 months
  presence of plaque (P) was evaluated as present/absent at six points of each tooth and recorded as percentages. Surgical site measurements were repeated at 3-and 6 months.
Bleeding on probing (BoP) | Baseline - 3months - 6 months
  Bleeding on probing (BoP) was evaluated as present/absent at six points of each tooth and recorded as percentages. Surgical site measurements were repeated at 3-and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Sadiye Gunpinar, Assoc. Prof., Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and statistical analysis plan.
Supporting Information: Study Protocol, SAP
Time Frame: Following the article publication of study protocol in a journal.
Access Criteria: The required data can be shared by responsible person (principal investigator of the study) upon reasonable request.